CLINICAL TRIAL: NCT05475977
Title: Role of Multislice Computed Tomography (MSCT) Chest in Differentiation Between Chronic Obstructive Pulmonary Disease(COPD) Patients According to Their Smoking Status
Brief Title: Role of MSCT of Chest in Differentiation Between COPD Patients According to Their Smoking Status
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Somaia Ahmad AbdAllah Ahmad (Other)
Responsible Party: Sponsor-Investigator, Somaia Ahmad AbdAllah Ahmad, Main investigator, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Somaia Ahmad
Record Dates: First submitted 2022-06-28; First posted 2022-07-27 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-08

CONDITIONS: Patient Participation
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- First Group: Thirty patients of COPD smokers patients.
  Interventions: Diagnostic Test: MSCT chest
- Second group: Thirty patients of COPD ex-smokers patients.
  Interventions: Diagnostic Test: MSCT chest
- Third group: Thirty patients of COPD non-smokers patients.
  Interventions: Diagnostic Test: MSCT chest

INTERVENTIONS:
Diagnostic Test: MSCT chest — Multi slice Computed Tomography of the chest

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a major cause of morbidity and mortality all over the world. Smoking is considered as an important risk factor, but other risk factors are present. Around 30 % of patients with COPD are non-smokers.

Cessation of smoking in patients with COPD causes decreases the presence of micronodules and other criteria of CT chest.

In last few years, some researchers reported that cessation of smoking raise the apparent extent of emphysema. The cause is not obvious, but this paradoxical fall in lung density is thaught to be resulting from decrease in inflammation after smoking cessation.

CT chest criteria of COPD in active smokers, non-smokers and ex-smokers seem to be different.

So, comparison between CT chest Criteria of COPD in smokers, ex-smokers and non-smokers will be searched in this study to detect the role of multislice computed tomography (MSCT) chest in differentiation between COPD patients according to their smoking status.

DETAILED DESCRIPTION:
Basic ethical principles of medical research; beneficence (do well), non-maleficence (do no harm), respect and distributive justice were implemented. The study will be carried out in accordance with the Declaration of Helsinki and the principles of good clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. All patients with chronic obstructive Pulmonary Disease.
2. Patients above 18 years.

Exclusion Criteria:

1. Patients with unclear smoking history.
2. Patients with active pneumonia.
3. Patients with acute COPD exacerbation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients either smokers, ex-smokers or non-smokers
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants with criteria of severe COPD | 18 months
  Criteria of severe COPD include emphysematous bullae, thick bronchial walls.

CONTACTS AND LOCATIONS:
Overall Officials: Somaia Ahmad AbdAllah Ahmad, M.B.B.Ch, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: Yes
COPD MSCT criteria smoking status
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2 years
Access Criteria: Medical researchers